CLINICAL TRIAL: NCT01978938
Title: A Phase 3, Randomized, Double-blind, Double-dummy, Multicenter, Prospective Study to Assess the Efficacy and Safety of Eravacycline Compared With Levofloxacin in Complicated Urinary Tract Infections
Brief Title: Efficacy and Safety Study of Eravacycline Compared With Levofloxacin in Complicated Urinary Tract Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TP-434-010
Record Dates: First submitted 2013-10-28; First posted 2013-11-08 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: cUTI
MeSH Terms: interventions — eravacycline; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Except for the responsible study site pharmacist or designee and separate unblinded clinical research associates to monitor drug supply and adherence to study drug blinding and randomization procedures, all study staff and participants were blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eravacycline (Experimental): Eravacycline was administered IV at a dose of 1.5 mg per kilogram (kg) of body weight every 24 hours (q24h). At minimum, the first 3 doses were administered IV. After an IV-to-PO transition, provided adequate clinical improvement, participants were administered 200 mg PO twice a day for a total therapy of 7 dosing cycles.
  Interventions: Drug: Eravacycline
- Levofloxacin (Active Comparator): Levofloxacin (750 mg) was administered IV q24h. At minimum, the first 3 doses were administered IV. After an IV-to-PO transition, provided adequate clinical improvement, participants were administered 750 mg PO once a day for a total therapy of 7 dosing cycles.
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Eravacycline
  Other Names: TP-434
  Arms: Eravacycline
Drug: Levofloxacin
  Other Names: Levaquin
  Arms: Levofloxacin

SUMMARY:
This is a phase 3, randomized, double-blind, double-dummy, multicenter, prospective study to assess the efficacy and safety of eravacycline compared with levofloxacin in participants with complicated urinary tract infections (cUTI).

DETAILED DESCRIPTION:
This study began with a 3-arm Lead-in portion to determine the oral (PO) dosing (200 or 250 milligrams [mg]) of eravacycline to be used with intravenously (IV) administered eravacycline for the Pivotal portion (2 arms). A PO dose of 200 mg was selected based on the unblinded Lead-in analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants with either:

a. Pyelonephritis and normal urinary tract anatomy (approximately 50% of the total population), OR b. cUTI with at least 1 of the following conditions associated with a risk for developing cUTI: i. Indwelling urinary catheter ii. Urinary retention (approximately 100 milliliters of residual urine after voiding) iii. Neurogenic bladder iv. Partial obstructive uropathy (such as, nephrolithiasis, bladder stones, and ureteral strictures) v. Azotemia of renal origin (not congestive heart failure or volume related) such that the serum blood urea nitrogen (BUN) is elevated (>20 mg/deciliters) AND the serum BUN: creatinine ratio is <15 vi. Surgically modified or abnormal urinary tract anatomy (such as, bladder diverticula, redundant urine collection system) EXCEPT surgery within the last month

Exclusion Criteria:

1. Concurrent use of non-study antibacterial drug therapy that would have a potential effect on outcome evaluations in participants with cUTI, including:

1. Participants with a history of a levofloxacin-resistant urinary tract infection
2. Likely to receive ongoing antibacterial drug prophylaxis prior to the late Post-Treatment visit (such as, participants with vesiculo-ureteral reflux)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2015-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (99):
- United States (6):
  - San Diego Clinical Trials, San Diego, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Tampa General Hospital, Tampa, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Sunrise Hospital and Medical Centre, Las Vegas, Nevada
  - Columbus Regional Research Institute, Columbus, Ohio
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment "Dr. Tota Venkova", Gabrovo, Department of Nephrology, Gabrovo
  - Multiprofile Hospital for Active Treatment "Dr. Stamen Iliev", Montana, Department of Nephrology and Dialysis, Montana
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski", Pleven, Urology Clinic, Pleven
  - Multiprofile Hospital for Active Treatment, Ruse, Department of Urology, Rousse
  - Multiprofile Hospital for Active Treatment, Sofia at Military Medical Academy, General Urology Clinic, Sofia
  - University Multiprofile Hospital for Active Treatment "Aleksandrovska", Sofia, Department of Laparoscopic Urology, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov", Sofia, Urology Clinic, Sofia
  - Multiprofile Regional Hospital for Active Treatment "Dr. Stefan Cherkezov", Veliko Tarnovo, Department of Urology, Veliko Tarnovo
- Colombia (2):
  - Fundacion Cardiomet, Armenia
  - De la Costa Clinic. Ltd. Research Centre, Barranquilla
- Czechia (5):
  - University Hospital Brno, Clinic of Urology, Brno
  - University Hospital Hradec Kralove, Clinic of Urology, Hradec Králové
  - Hospital Novy Jicin, Department of Urology, Nový Jičín
  - University Hospital Olomouc, Olomouc
  - Thomayer Hospital, Department of Urology, Prague
- Estonia (4):
  - East Viru Central Hospital, Surgery Clinic, Kohtla-Järve
  - East Tallinn Central Hospital, Department of Internal Medicine, Tallinn
  - West Tallinn Central Hospital, Department of Urology, Tallinn
  - Tartu University Hospital, Surgery Clinic, Department of Urology and Renal Transplantation, Tartu
- Georgia (5):
  - Western Georgia National Medical Center, Kutaisi
  - Aversi Clinic, Tbilisi
  - Modern Medical Technologies - Guram Karazanashvili's clinic, Tbilisi
  - Research Institute of Clinical Medicine, Tbilisi
  - Tsulukidze National Center of Urology, Tbilisi
- Greece (2):
  - Evaggelismos Hospital, Kolonaki
  - Papageorgiou General Hospital, Thessaloniki
- Hungary (6):
  - Principal SMO Kft., Baja
  - Jahn Ferenc South Pest Hospital, Department of Urology, Budapest
  - Petz Aladar County Teaching Hospital, Department of Urology, Győr
  - Elisabeth Teaching Hospital and Rehabilitation Institute of Sopron, Department of Urology, Sopron
  - Csongrad County Dr. Bugyi Istvan Hospital, Department of Urology, Szentes
  - St. Borbala Hospital, Department of Urology, Tatabánya
- Zion Medical Center, Haifa, Israel
- Hospital Mater Domini, Castellanza, Italy
- Latvia (5):
  - Liepajas Regional Hospital, Liepāja
  - P. Stradins Clinical University Hospital, Riga
  - Riga East University Hospital, LLC, Riga
  - SIA 'URO' Clinic, Riga
  - Vidzemes Hospital, Valmiera
- Mexico (2):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara
  - Hospital Civil Guadalajara Dr. Juan I. Mendoza, Guadalajara
- Moldova (2):
  - National Scientific Practical Center for Emergency Medicine, Department of Urology, Chisinau
  - Republican Clinical Hospital, Department of Urology, Chisinau
- Poland (5):
  - Boni Fratres Catoviensis Sp. z o.o., Department of Internal Diseases with Cardiologic Diagnostics Unit, Katowice
  - Military Medical Academy University Teaching Hospital - Central Veterans' Hospital, Clinical and Didactic Center of the Medical University of Lodz, Teaching Department of Nephrology, Hypertension and Renal Transplantation, Lodz
  - Medicome Sp. z o.o., Oświęcim
  - HEUREKA Hanna Szalecka, Piaseczno
  - Pope John Paul 2nd Independent Public Provincial Hospital, Zamość
- Romania (7):
  - Emergency Clinical County Hospital Brasov, Brasov
  - "Prof. Dr. Th. Burghele" Clinical Hospital, Bucharest
  - Delta Hospital, Bucharest
  - Craiova Emergency Clinical County Hospital, Craiova
  - Clinical Hospital "Dr. C. I. Parhon", Iași
  - Oradea Clinical Municipal Hospital "Dr. Gavril Curteanu", Oradea
  - Sibiu County Emergency Clinical Hospital, Sibiu
- Russia (16):
  - Central Clinical Hospital of Civil Aviation, Moscow
  - City Clinical Hospital #57 under Moscow Healthcare Department, Moscow
  - Federal Clinical Center for High Medical Technologies, Moscow
  - City Clinical Hospital of Emergency Care #2, Novosibirsk
  - Penza Regional Clinical Hospital n.a. N.N. Burdenko, Penza
  - Rostov State Medical University, Rostov-on-Don
  - North-Western State Medical University n.a. I.I. Mechnikov, Saint Petersburg
  - Saint-Petersburg Scientific Research Institute for Phthisiopulmonology, Saint Petersburg
  - St. Petersburg Clinical Hospital under the Russian Academy of Sciences, Saint Petersburg
  - St. Petersburg State Healthcare Institution: City Hospital #15, Saint Petersburg
  - St. Petersburg State Healthcare Institution: St. George the Martyr City Hospital, Saint Petersburg
  - St. Petersburg State-Funded Healthcare Institution: City Hospital #26, Saint Petersburg
  - Saratov State Medical University n.a. V.I. Razumovsky, Saratov
  - Smolensk Regional Clinical Hospital, Smolensk
  - Novgorod Regional Clinical Hospital, Veliky Novgorod
  - Vsevolozhsk Clinical Central District Hospital, Vsevolozhsk
- South Africa (4):
  - Lakeview Hospital, Benoni
  - Clinresco Centres, Kempton Park
  - Mzansi Ethical Research Centre, Middleburg
  - St. Georges Hospital, Port Elizabeth
- Ukraine (18):
  - Regional Municipal Institution "Chernivtsi Regional Hospital", Chernivtsi
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Dnipropetrovsk
  - Dnipropetrovsk I.I. Mechnikov Regional Clinical Hospital, Dnipropetrovsk
  - Ivano-Frankivsk City Clinical Hospital #1, Ivano-Frankivsk
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - O.I. Meschaninov Clinical Hospital of Emergency and Urgent Medical Care, Kharkiv
  - Shapoval Regional Clinical Center of Urology and Nephrology, Kharkiv
  - Khmelnytskyi Regional Hospital, Khmelnytskyi
  - Institute of Urology, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Lviv Regional Clinical Hospital, Lviv
  - Mykolaiv Regional Hospital, Center for Nephrology and Dialysis, Mykolaiv
  - City Clinical Hospital #10, Urology Department #1, Odesa
  - Odesa Regional Clinical Hospital, Odesa
  - Poltava M.V. Sklifosovskyi Regional Clinical Hospital, Poltava
  - State Institution: Uzhhorod Railway Station Clinical Hospital under State Territorial Industry-Specific Association:Lviv Railway, Uzhhorod
  - Vinnytsia M.I. Pyrohov Regional Clinical Hospital, Vinnytsia
  - Municipal Institution "Zaporizhzhia Reqional Clinical Hospital" of Zaporizhzhia Regional Councill, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of complicated urinary tract infection (cUTI), including participants with acute pyelonephritis, were recruited into this study.
Pre-assignment Details: Screening and baseline assessments were performed after informed consent was obtained and within 36 hours prior to enrollment.
Groups:
- Eravacycline: Eravacycline was administered intravenously (IV) at a dose of 1.5 milligrams per kilogram (mg/kg) of body weight every 24 hours (q24h). At minimum, the first 3 doses were administered IV. After an IV-to-oral (PO) transition, provided adequate clinical improvement, participants were administered 200 mg PO twice a day (BID) for a total therapy of 7 dosing cycles.
- Levofloxacin: Levofloxacin (750 mg) was administered IV q24h. At minimum, the first 3 doses were administered IV. After an IV-to-PO transition, provided adequate clinical improvement, participants were administered 750 mg PO once a day (QD) for a total therapy of 7 dosing cycles.
Period: Overall Study
Arm/Group | Eravacycline | Levofloxacin
Started | 455 | 453
Received at Least 1 Dose of Study Drug (1 participant in the eravacycline group and 2 in the levofloxacin group did not receive study drug.) | 454 | 451
Completed | 432 | 439
Not Completed | 23 | 14
Not completed — Lost to Follow-up | 12 | 6
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Adverse Event, non-fatal | 2 | 1
Not completed — Participant noncompliance | 1 | 1
Not completed — Did not meet inclusion criteria | 0 | 1
Not completed — Previously scheduled procedure | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all randomized participants regardless of whether or not the participant received study drug.
Groups:
- Eravacycline: Eravacycline was administered IV at a dose of 1.5 mg/kg of body weight q24h. At minimum, the first 3 doses were administered IV. After an IV-to-PO transition, provided adequate clinical improvement, participants were administered 200 mg PO BID for a total therapy of 7 dosing cycles.
- Levofloxacin: Levofloxacin (750 mg) was administered IV q24h. At minimum, the first 3 doses were administered IV. After an IV-to-PO transition, provided adequate clinical improvement, participants were administered 750 mg PO QD for a total therapy of 7 dosing cycles.
- Total: Total of all reporting groups
Arm/Group | Eravacycline | Levofloxacin | Total
Number analyzed (Participants) | 455 | 453 | 908
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 291 | 301 | 592
  >=65 years | 164 | 152 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (18.82) | 51.7 (19.81) | 52.7 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 302 | 593
  Male | 164 | 151 | 315

OUTCOME MEASURES:

1. Primary Outcome: Participants In The Microbiological Intent-To-Treat (Micro-ITT) Population With A Responder Outcome At The Post-Treatment (PT) Visit
Description: This was the primary outcome measure for the Food and Drug Administration (FDA). The primary objective was to demonstrate the non-inferiority (NI) of eravacycline to levofloxacin in responder outcome, which was derived from both clinical and microbiological responses, in the micro-ITT population. Clinical responses were either cure, failure, or indeterminate/missing; microbiological responses were characterized programmatically as either success, failure, or indeterminate/missing. Clinical cure was defined as complete resolution or significant improvement of signs or symptoms of the infection; microbiological success was a reduction of the baseline pathogen(s) to <10^4 colony-forming units/milliliter (CFU/mL). An outcome of Responder required a clinical response of cure and a microbiological response of success. Any other combination of the clinical and microbiological responses was considered either Non-responder or Indeterminate.
Time Frame: PT Visit
Population: micro-ITT included all participants in the ITT population who had at least 1 baseline bacterial pathogen from a urine or blood culture that caused a urinary tract infection (UTI) against which eravacycline had expected antibacterial activity. ITT included all randomized participants, regardless of receiving study drug or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Eravacycline | Levofloxacin
Number analyzed (Participants) | 298 | 302
Participants
  Responder | 180 | 202
  Non-responder | 100 | 91
  Indeterminate | 18 | 9
Statistical Analysis 1: Comparison: Eravacycline vs Levofloxacin; For the FDA, an NI margin of 10% was used, which was based on historical data regarding the treatment effect of antibiotics. A 10% NI margin for the Responder outcome is robust and can sufficiently confirm a clinically meaningful treatment effect of eravacycline in the treatment of cUTI; Test type: Non-Inferiority — The NI test was based on the lower limit of the 2-sided 95% confidence interval (CI), using the method proposed without stratification by Miettinen and Nurminen. If the lower limit of the 95% CI for the difference in Responder (clinical cure and microbiologic success) rates in the micro-ITT population exceeded -10%, then the null hypothesis was rejected and the NI of eravacycline to levofloxacin was declared; Treatment Difference = -6.5, 95% CI 2-sided [-14.1 to 1.2]

2. Secondary Outcome: Participants In The Microbiological Modified ITT (Micro-MITT) Population With A Microbiological Response
Description: This outcome measure (FDA and the European Medicines Agency [EMA]) compared the microbiological responses of eravacycline to levofloxacin for both treatment groups in the micro-MITT population. Responses were success, failure, or indeterminate/missing. Success was considered a reduction of the baseline pathogen(s) to <10^4 CFU/mL. Failure required blood cultures at or beyond end of therapy (EOT) to be positive for baseline pathogen(s), or urine culture to grow ≥10^4 CFU/mL of the baseline pathogen(s). Indeterminate/missing indicated no interpretable culture data available.
Time Frame: PT Visit
Population: micro-MITT included all micro-ITT participants who received ≥1 dose of study drug. micro-ITT: all ITT participants with ≥1 baseline bacterial pathogen from a urine or blood culture that caused a UTI against which eravacycline had expected antibacterial activity. ITT: all randomized participants, regardless of receiving study drug or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Eravacycline | Levofloxacin
Number analyzed (Participants) | 297 | 302
Participants
  Success | 194 | 213
  Failure | 85 | 78
  Indeterminate/missing | 18 | 11

3. Secondary Outcome: Participants In The Microbiologically Evaluable (ME) Population With A Microbiological Response
Description: This outcome measure (FDA and EMA) compared the microbiological responses of eravacycline to levofloxacin for both treatment groups in the ME population. Responses were either success or failure. Indeterminate/missing responses were not included. Success was considered a reduction of the baseline pathogen(s) to <10^4 CFU/mL. Failure required blood cultures at or beyond EOT to be positive for baseline pathogen(s), or urine culture to grow ≥10^4 CFU/mL of the baseline pathogen(s). Indeterminate/missing indicated no interpretable culture data available. Populations: ME, all micro-ITT and clinically-evaluable (CE) participants with a suitable urine specimen and an interpretable urine culture; micro-ITT, all participants with ≥1 baseline bacterial pathogen from a urine or blood culture that caused a UTI against which eravacycline had expected antibacterial activity; ITT, all randomized participants, regardless of receiving study drug or not.
Time Frame: PT Visit
Population: ME: all micro-ITT and CE participants with a suitable urine specimen and an interpretable urine culture. CE: all randomized participants dosed with no other antimicrobials (unless allowed by protocol), had an investigator clinical response assessment of "success" or "failure" at the assessment visit, and had no other major protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | Eravacycline | Levofloxacin
Number analyzed (Participants) | 255 | 276
Participants
  Success | 180 | 203
  Failure | 75 | 73

ADVERSE EVENTS:
Time Frame: The time frame for adverse event reporting was from the first dose of study drug through 30 days after the last dose of study drug or the late post-treatment visit (whichever was later).
Description: The safety population was all randomized subjects who receive any amount of study drug. All safety analyses were conducted in this population and are presented by treatment actually received (not as randomized). One subject was randomized to levofloxacin but received eravacycline, therefore Eravacycline N = 455; Levofloxacin N= 450
Arm/Group | Eravacycline | Levofloxacin
All-Cause Mortality (participants affected / at risk) | 1/455 | 0/450
Serious Adverse Events (participants affected / at risk) | 7/455 | 6/450
Other Adverse Events (participants affected / at risk) | 129/455 | 26/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eravacycline (N=455) | Levofloxacin (N=450)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eravacycline (N=455) | Levofloxacin (N=450)
Nausea (Gastrointestinal disorders) | 82 | 14
Vomiting (Gastrointestinal disorders) | 33 | 6
Headache (Nervous system disorders) | 14 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications should include input from the PI, his/her colleagues, other PIs in this trial and the Sponsor's personnel; such input should be reflected in the authorship. Agreement of order of authors should be established before writing a manuscript. The PI interested in participating in writing the manuscript should contact the Sponsor. The PI shall not make any publication without the Sponsor's prior written approval, which may be withheld or granted by the Sponsor, in its sole discretion.